CLINICAL TRIAL: NCT06021808
Title: Epicardial Left Atrial Appendage Clipping Versus Novel Oral Anticoagulants to Reduce Stroke Risk in Non-paroxysmal Atrial Fibrillation: a Multicenter Randomized Controlled Trial
Brief Title: LAA Clipping Versus NOACs to Prevent Stroke in Non-paroxysmal Atrial Fibrillation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-2059
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Non-paroxysmal Atrial Fibrillation
Keywords: left atrial appendage clipping; Stroke; Oral anticoagulation; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAA clipping group (Experimental): In this arm, participants are performed thoracoscopic LAA clipping.
  Interventions: Procedure: Thoracoscopic LAA clipping
- NOACs group (Active Comparator): Patients randomized to NOAC therapy will begin long-term oral administration of NOACs immediately after enrollment.
  Interventions: Drug: Novel oral anticoagulant

INTERVENTIONS:
Procedure: Thoracoscopic LAA clipping — The surgeons measured the length of the base of the LAA, an appropriately sized LAA clip is then inserted with the aid of a thoracoscope and placed parallel to the base of the LAA.
  Arms: LAA clipping group
Drug: Novel oral anticoagulant — For patients with creatinine clearance ≥50 ml/min, oral rivaroxaban 20 mg daily was administered, whereas for patients with creatinine clearance between 30-49 ml/min, oral rivaroxaban 15 mg daily was administered.
  Arms: NOACs group

SUMMARY:
This trial is designed to examine the hypothesis that thoracoscopic LAA clipping is superior to NOACs for stroke, systemic embolism, all-cause mortality, major bleeding events and clinically relevant nonmajor bleeding events in AF patients at high risk of embolism (CHA2DS2-VASc ≥2 in men and ≥3 in women) that are not undergoing ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most prevalent cardiac arrhythmia disease, and the incidence of AF increases markedly with age and approximately doubles with each decade. According to the previous study, the incidence of stroke were five times in patients with AF than those in the general population. Systemic oral anticoagulant is a well-established, guideline-recommended therapy for the prevention of ischemic stroke in patients with nonvalvular AF at high risk of embolism (CHA2DS2-VASc scores ≥2 in men and ≥3 in women), and the guidelines recommend that the novel oral anticoagulants (NOACs) be preferred (Class I, Level of evidence A). However, a significant proportion of patients with nonvalvular AF have difficulties in long-term oral anticoagulant therapy, due to medication adherence and contraindications to oral anticoagulants. Also, several randomized controlled trials indicated that bleeding risk remained high with novel oral anticoagulants. Therefore, it is essential to explore alternative treatment strategies for stroke prevention in patients with nonvalvular AF.

It has been reported that the left atrial appendage (LAA) is suspected as a vital source of cerebral emboli and may lead to ischemic stroke, removal or closure of the LAA may be an alternative to oral anticoagulants. Various surgical or interventional approaches have been developed to close or occlude LAA to prevent stroke in AF patients, such as percutaneous LAA occlusion, suture ligation, and surgical excision. However, these techniques suffer from incomplete LAA closure or the presence of residual blood flow, which can lead to thrombosis and stroke. Thoracoscopic LAA clip, on the other hand, cloud block blood flow between the LAA and the left atrium (LA), achieving isolation of LAA and preventing thrombi and strokes. A previous study has demonstrated a high 95% success rate of LAA clipping without operation-related complications, and freedom from stroke was 99.1% at a median follow-up of 20 months. Therefore, LAA clipping is an effective and durable method in stroke prevention. However, currently high-quality RCTs are lacking to support the superiority of LAA clipping compared with NOACs in terms of stroke prevention and safety. In this trial, the investigators designed a multicenter prospective RCT to compare the efficacy and safety of thoracoscopic LAA clipping and NOACs in patients with non-paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Persistent or long-standing persistent AF documented by medical history or direct electrocardiogram.
* CHA2DS2-VASc ≥2 in men and ≥3 in women.
* Agree to perform thoracoscopic LAA occlusion procedure.

Exclusion Criteria:

* With electrical cardioversion or ablation intent.
* Other heart diseases with surgical indications.
* Ischemic stroke and other cardiac embolic events within 30 days.
* Major clinical bleeding event within 30 days.
* Contraindications to anticoagulation.
* Intracardiac thrombus.
* Left ventricular ejection fraction (LVEF) < 30%.
* Active systemic infection or infective endocarditis or pericarditis
* Severe liver disease (acute clinical hepatitis, chronic active hepatitis, cirrhosis) or alanine transaminase (ALT)/ aspartate transaminase (AST) greater than 3 times the upper limit of normal value.
* Severe renal insufficiency (eGFR ≤ 30mL/min).
* Other diseases requiring oral anticoagulants.
* Active aortic plaque.
* Acute coronary syndrome within 3 months.
* Symptomatic carotid artery stenosis.
* Patients requiring dual antiplatelet drug therapy.
* Previous cardiac and left lung surgery.
* Severe left pleural and pericardial adhesions.
* Pregnant or breastfeeding patients.
* Metal allergies.
* Terminal illness with a life expectancy of less than 2 years.
* Participation in other clinical studies at the time of enrollment.
* Refuse to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Rate of composite endpoint | At 24-month after intervention
  Stroke, systemic embolism, all-cause mortality, major bleeding event, and clinically relevant non-major bleeding event.

SECONDARY OUTCOMES:
Rate of stroke | At 24-month after intervention
  Acute episodes of focal or global neurological dysfunction due to cerebral, spinal cord or retinal vascular injury from haemorrhage or infarction. Symptoms or signs must have lasted ≥ 24 hours, or symptoms/signs may have lasted less than 24 hours if demonstrated by CT, MRI, or autopsy.
Rate of systemic embolism | At 24-month after intervention
  Confirmed by imaging or angiography
Rate of all-cause mortality | At 24-month after intervention
  Deaths from all causes
Rate of major bleeding event | At 24-month after intervention
  1. fatal haemorrhage, and/or
  2. Symptomatic haemorrhage in a critical area or organ, such as intracranial, intravertebral, intraocular, retroperitoneal, intra-articular or intrapericardial, or intramuscular haemorrhage leading to osteofascial compartment syndrome, and/or 3. haemorrhage that results in a fall in haemoglobin level of 2.0 g/dL or more, or that results in the importation of two or more units of whole blood or red blood cells.
Rate of clinically relevant non-major bleeding event | At 24-month after intervention
  Bleeding events that do not meet the criteria for an ISTH major bleeding event but requires hospitalisation or a change in antithrombotic treatment strategy or requires invasive management.
Rate of surgery-related complications | At 24-month after intervention
  Incidence of in-hospital death, in-hospital stroke, intermediate small-incision open thoracotomy or median open thoracotomy, and postoperative re-intervention due to hemorrhage, pneumothorax, and pyothorax.
Rate of minor bleeding events | At 24-month after intervention
  Bleeding events that do not meet the ISTH criteria for a major bleeding event, do not meet the criteria for a clinically relevant non-major bleeding event, and do not require the subject to seek additional assistance from medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD,PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu C, Li H, Lei C, Wang Y, Chen S, Zhao Y, Zheng Z. Epicardial left atrial appendage clipping versus direct oral anticoagulant to reduce stroke risk in non-paroxysmal atrial fibrillation (LAA-CLIP): rationale, design and study protocol for a multicentre randomised controlled trial. BMJ Open. 2024 Mar 5;14(3):e083153. doi: 10.1136/bmjopen-2023-083153. PMID 38448081